CLINICAL TRIAL: NCT02082106
Title: Metabolic and Physiological Stress During Alpine Skiing, Cross-country Skiing and Indoor Training in Untrained and Trained Persons.
Brief Title: Metabolic and Physiological Stress During Skiing.
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Head of Institute; University Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University
Other Study IDs: UISM-2014-MET-SKI
Record Dates: First submitted 2014-02-11; First posted 2014-03-10 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: alpine skiing; cross country skiing; indoor cycling; physical fitness; training status; metabolic equivalent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood serum, blood plasma, blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- males/females: Participants should be capable of alpine skiing and cross country skiing.
  Interventions: Other: Alpine skiing; Other: cross country skiing; Other: Indoor training (cycling)

INTERVENTIONS:
Other: Alpine skiing
Other: cross country skiing
Other: Indoor training (cycling)

SUMMARY:
Problem description In industrialized countries there is a rapid increase in the number of senior citizens. In Austria more than 50% of the population is overweight, with highest prevalence in the age group from 60 to 74 yrs and the WHO lists physical inactivity as one of the main behavioral risk factors of cardiovascular diseases.

Especially in winter months, activity related energy expenditure was 40% and 31% lower in the US and Canada, respectively. In addition, in an Austrian study the winter season was associated with higher blood pressure, total cholesterol and body mass index, giving an increasing risk of chronic coronary disease by 6.8% in men and 3.6% in women.

Therefore, the development of intervention programs that overcome the winter physical activity deficit and be feasible also for elderly should be goal of future research. Alpine skiing (AS) and cross country skiing (XCS) have a long standing tradition in Austria and could potentially fill the winter physical activity gap. The Salzburg Skiing for the Elderly Study (SASES) has found AS to be a save and feasible possibility to improve the health of the aged population in many parameters. XCS as a competitive sport is already well explored but there are hardly any studies about its effects in the normal or elderly population. Unfortunately knowledge about the differences between AS and XCS in the physiological adaptation processes in the elderly population is also lacking.

Aims and hypotheses of the pre-study In order to standardize training interventions, the present pre-study aims at comparing physiological and metabolic parameters between AS, XCS and IT. Therefore, the results of the pre-study serve as determinants for the training parameters of the above mentioned main study.

We postulate that, based on the results of the present study, it is possible to set up comparable isocaloric training sessions for AS, XCS and IT for elderly and unfit persons.

Furthermore, we assume that elderly and unfit subjects are able to perform a full spectrum of intensities and techniques necessary to set appropriate stimuli for isocaloric comparison.

We hypothesize arterial stiffness indices and circulating microRNA (miRNA) patterns to change due to one bout of physical activity of AS, XCS, and IT with variations depending on the kind of sport.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* male or female
* age: 30+ years
* inconspicuous ECG
* Non-smoker for at least one year
* proper skills in alpine skiing and cross-country skiing

Exclusion Criteria:

* Participation in other clinical trials at the same time or within the previous 6 months
* Tiffeneau-Pinelli index: Forced Expiratory Volume in first second (FEV1) / Forced Vital Capacity (FVC) <60% with/without symptoms (coughing, sputum) or other evidence of a pulmonary disease
* medical condition which conflicts with participation in training
* Intake of anticoagulants
* Alcohol or drug abuse
* Severe obesity: BMI >40

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty healthy subjects (male=10/female=10) aged 30+ will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption (VO2) | 12 weeks
  VO2 will be measured during during physical examination, indoor training, Alpine Skiing, and Cross Country Skiing. VO2 will be transformed into metabolic equivalents to calculate isocaloric training parameters for the different kind of sport.

SECONDARY OUTCOMES:
Pulse wave analysis (PWA) | 12 weeks
  PWA will be measured before/after physical examination, indoor training, Alpine Skiing, and Cross Country Skiing. PWA will be done by oscillometric measurement to calculate influence of acute exercise and training status on several pulse wave parameters.

OTHER OUTCOMES:
RNA | 12 weeks
  Total RNA will be isolated from stored plasma and blood cell samples. All samples will be screened for influence of acute exercise (before/after physical examination and indoor training).
Nitric oxide (NO) | 12 weeks
  NO will be quantified out of stored blood samples and serves as a possible surrogate parameter of pulse wave analysis.
Metabolic screening | 12 weeks
  Metabolic parameters (e.g. glucose, lactate) will be quantified out of stored blood samples: These parameters serve as determinants of the different exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Josef Niebauer, MBA, Prof. Dr.Dr., Principal Investigator — Paracelsus Medical University; Martin Schoenfelder, Dr., Study Chair — Research Institute of Moleclar Sport and Rehabilitation Medicine, Paracelsus Medical University Salzburg, Austria; Thomas Stoeggl, Prof. Dr., Study Chair — Department of Sport Sciency and Kinesiology - University of Salzburg
Locations (1):
- University Institute of Sports Medicine, Prevention and Rehabilitation, Salzburg, Austria

REFERENCES:
- [Background] Muller E, Gimpl M, Poetzelsberger B, Finkenzeller T, Scheiber P. Salzburg Skiing for the Elderly Study: study design and intervention--health benefit of alpine skiing for elderly. Scand J Med Sci Sports. 2011 Aug;21 Suppl 1:1-8. doi: 10.1111/j.1600-0838.2011.01336.x. PMID 21679318
- [Background] Niederseer D, Ledl-Kurkowski E, Kvita K, Patsch W, Dela F, Mueller E, Niebauer J. Salzburg Skiing for the Elderly Study: changes in cardiovascular risk factors through skiing in the elderly. Scand J Med Sci Sports. 2011 Aug;21 Suppl 1:47-55. doi: 10.1111/j.1600-0838.2011.01341.x. PMID 21679323
- [Background] Muller E, Gimpl M, Kirchner S, Kroll J, Jahnel R, Niebauer J, Niederseer D, Scheiber P. Salzburg Skiing for the Elderly Study: influence of alpine skiing on aerobic capacity, strength, power, and balance. Scand J Med Sci Sports. 2011 Aug;21 Suppl 1:9-22. doi: 10.1111/j.1600-0838.2011.01337.x. PMID 21679319
- [Background] Finkenzeller T, Muller E, Wurth S, Amesberger G. Does a skiing intervention influence the psycho-social characteristics of the elderly? Scand J Med Sci Sports. 2011 Aug;21 Suppl 1:69-75. doi: 10.1111/j.1600-0838.2011.01344.x. PMID 21679326
- See also: Research Institute of Molecular Sport and Rehabilitation Medicine — http://www.pmu.ac.at/mol-sportmed.html
- See also: University Institute of Sports Medicine, Prevention and Rehabilitation — http://www.salk.at/sportmedizin.html